CLINICAL TRIAL: NCT06958172
Title: Investigation of The Effects of Core Stabilization, Hip and Thoracic Mobility Exercises on Desk Workers With Postural Disorders
Brief Title: The Effects of Core Stabilization on Desk Workers With Postural Disorders
Acronym: CORE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Collaborators: Istinye University (Other)
Responsible Party: Principal Investigator, Muhammed ARCA, Director, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Istinye University
Record Dates: First submitted 2025-03-13; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Postural Imbalance; Worker Health
Keywords: Balance; Core Stabilization; Mobility Exercise
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): only performed the same home exercise program
- Other (Experimental): Exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Study Group received core stabilization, thoracic mobility and hip mobility exercises
  Arms: Other

SUMMARY:
This study aimed to investigate the effects of core, thoracic and hip mobility exercises on trunk stabilization and postural improvement in desk workers with postural disorders.

DETAILED DESCRIPTION:
A randomized controlled study was conducted with 40 desk workers aged 25-45. Participants were divided into two groups: Study Group (n=21) and Control Group (n=20). Participants in the Study Group received core stabilization, thoracic Participants in the Control Group performed mobility and hip mobility exercises, while participants in the Control Group only performed the same home exercise program. Before and after treatment, trunk stabilization of the participants was evaluated with the Plank test and Sorenson test, and their balance was evaluated with the Y balance test .

ELIGIBILITY:
Inclusion Criteria:

* Having a desk job
* Being between the ages of 25-45,
* Written approval of participation in the study by himself/herself or his/her legal representative

Exclusion Criteria:

* Having had surgery within the last six months,
* Having a previously identified and diagnosed cardiovascular or pulmonary disease

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Assessment Methods | 2 months
  Participants' trunk stabilization with Plank-Sorenson and Y Balance Test will be assessed before and after treatment.
Plank test and Sorenson test | 2 months
  It is one of the basic static tests used to measure trunk endurance. Subjects are asked to lie face down, stand on their toes with their forearms and elbows shoulder-width apart and their pelvis lifted, and their neck, shoulders, back, hips and legs forming a straight line parallel to the ground, and the subject is asked to maintain this posture. The time until the subject gets tired and/or breaks their posture is recorded in seconds from the start of the time
Y balance test | 2 months
  Y Balance Test" platform was used to measure dynamic postural control . The leg length of each participant was measured in centimeters in the supine position bilaterally and anteriorly. medial from superioriliac point Malleolus The measurements were recorded by measuring the distal part. The measurements were tested barefoot, in 3 directions, anterior (ANT) reach as the distance between the participant's central toe tip, and posterolateral (PL) and posteromedial (PM) reach as the farthest point from the heel. During the trial, the participants are asked to keep their hands on the iliac crest and their heels on the floor and to lightly touch the farthest point with the toe tip of the reaching foot. in order to eliminate the leg length advantage, the scores obtained were normalized using the formula "Best Reach Distance/Leg Length ) x100 = % maximum reach distance" for each direction

CONTACTS AND LOCATIONS:
Overall Officials: Mertcan Kızılpınar, Study Chair — İstinye University

IPD SHARING:
Plan to Share IPD: No
Due to confidentiality of patient data